CLINICAL TRIAL: NCT06921486
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase IIb/III Clinical Trial to Evaluate the Efficacy and Safety of Efsubaglutide Alfa Injection in Overweight and Obese Subjects
Brief Title: The Efficacy and Safety of Efsubaglutide Alfa Injection in Overweight and Obese Subjects (ENLIGHT)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Yinnuo Pharmaceutical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YN011-W303; YN011-W202 (Other: Guangzhou Innogen Pharmaceutical Group Co., Ltd.); YN011-W303 (Other: Guangzhou Innogen Pharmaceutical Group Co., Ltd.)
Record Dates: First submitted 2025-03-28; First posted 2025-04-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Phase IIb：Efsubaglutide Alfa 5 mg QW (Experimental): The drug is administered once weekly, starting with a titration dose of 1 mg. The dose is up-titrated every 2 weeks in the sequence of 1 mg → 5 mg, reaching the target dose of 5 mg at Week 3 (W3). From W3 to W18, the treatment is maintained at a 5 mg dose.
  Interventions: Drug: Phase IIb：Efsubaglutide Alfa 5 mg QW
- Phase IIb：Efsubaglutide Alfa 10 mg QW (Experimental): The drug is administered once weekly, starting with a titration dose of 1 mg. The dose is up-titrated every 2 weeks in the sequence of 1 mg → 5 mg → 10 mg, reaching the target dose of 10 mg at Week 5 (W5). From W5 to W18, the treatment is maintained at a 10 mg dose.
  Interventions: Drug: Phase IIb：Efsubaglutide Alfa 10 mg QW
- Phase IIb：Efsubaglutide Alfa 20 mg QW (Experimental): The drug is administered once weekly, starting with a titration dose of 1 mg. The dose is up-titrated every 2 weeks in the sequence of 1 mg → 5 mg → 10 mg → 20 mg, reaching the target dose of 20 mg at Week 7 (W7). From W7 to W18, the treatment is maintained at a 20 mg dose.
  Interventions: Drug: Phase IIb：Efsubaglutide Alfa 20 mg QW
- Phase IIb：Efsubaglutide Alfa 20 mg Q2W (Experimental): From Week 1 (W1) to Week 6 (W6), the drug is administered once weekly, starting with a titration dose of 1 mg. The dose is up-titrated every 2 weeks in the sequence of 1 mg → 5 mg → 10 mg → 20 mg, reaching the target dose of 20 mg at Week 7 (W7). From W7 to W18, the drug is administered every two weeks and maintained at a 20 mg dose.
  Interventions: Drug: Phase IIb：Efsubaglutide Alfa 20 mg Q2W
- Phase IIb：Placebo (Placebo Comparator): Once weekly
  Interventions: Drug: Phase IIb：Placebo
- Phase III：Recommended Phase 3 Dose (RP3D) Low Dose QW (Experimental): The drug is administered once weekly, starting with a titration dose of 1 mg. The dose is up-titrated every 2 weeks in the sequence of 1 mg → 5 mg → 10 mg → 20 mg, The dose escalation continues until reaching the RP3D Low Dose, and then the RP3D is maintained. The total cumulative duration of drug administration (from the first dose to the end of maintenance) is 48 weeks, with the once-weekly administration frequency retained throughout the entire period.
  Interventions: Drug: Phase III：Recommended Phase 3 Dose Low Dose
- Phase III：Recommended Phase 3 Dose (RP3D) High Dose QW (Experimental): The drug is administered once weekly, starting with a titration dose of 1 mg. The dose is up-titrated every 2 weeks in the sequence of 1 mg → 5 mg → 10 mg → 20 mg, The dose escalation continues until reaching the RP3D High Dose, and then the RP3D is maintained. The total cumulative duration of drug administration (from the first dose to the end of maintenance) is 48 weeks, with the once-weekly administration frequency retained throughout the entire period.
  Interventions: Drug: Phase III：Recommended Phase 3 Dose High Dose
- Phase III：Recommended Phase 3 Dose (RP3D) High Dose Q2W (Experimental): The drug is administered once weekly, starting with a titration dose of 1 mg. The dose is up-titrated every 2 weeks in the sequence: 1 mg → 5 mg → 10 mg → 20 mg. Dose escalation continues until reaching the RP3D High Dose. Once the RP3D High Dose is achieved, the treatment regimen transitions to alternating weekly between RP3D High Dose and placebo for the remainder of the study. The total cumulative duration of drug administration (from the first dose to the end of the maintenance phase) remains 48 weeks, with the once-weekly administration frequency retained throughout. Blinding is maintained across all treatment groups to ensure unbiased evaluation of efficacy and safety.
  Interventions: Drug: Phase III：Recommended Phase 3 Dose High Dose; Drug: Phase III：Placebo
- Phase III：Placebo (Placebo Comparator): Once weekly
  Interventions: Drug: Phase III：Placebo

INTERVENTIONS:
Drug: Phase IIb：Efsubaglutide Alfa 5 mg QW — IIb：Efsubaglutide Alfa 5 mg QW
  Arms: Phase IIb：Efsubaglutide Alfa 5 mg QW
Drug: Phase IIb：Efsubaglutide Alfa 10 mg QW — Efsubaglutide Alfa 10 mg QW
  Arms: Phase IIb：Efsubaglutide Alfa 10 mg QW
Drug: Phase IIb：Efsubaglutide Alfa 20 mg QW — Efsubaglutide Alfa 20 mg QW
  Arms: Phase IIb：Efsubaglutide Alfa 20 mg QW
Drug: Phase IIb：Efsubaglutide Alfa 20 mg Q2W — Efsubaglutide Alfa 20 mg Q2W
  Arms: Phase IIb：Efsubaglutide Alfa 20 mg Q2W
Drug: Phase IIb：Placebo — Placebo
  Arms: Phase IIb：Placebo
Drug: Phase III：Recommended Phase 3 Dose High Dose — The Recommended Phase 3 Dose High Dose confirmed by the IDMC (Independent Data Monitoring Committee) based on the safety and efficacy data results from the 18-week Phase IIb.
  Arms: Phase III：Recommended Phase 3 Dose (RP3D) High Dose Q2W; Phase III：Recommended Phase 3 Dose (RP3D) High Dose QW
Drug: Phase III：Recommended Phase 3 Dose Low Dose — The Recommended Phase 3 Dose Low Dose confirmed by the IDMC (Independent Data Monitoring Committee) based on the safety and efficacy data results from the 18-week Phase IIb.
  Arms: Phase III：Recommended Phase 3 Dose (RP3D) Low Dose QW
Drug: Phase III：Placebo — Placebo
  Arms: Phase III：Placebo; Phase III：Recommended Phase 3 Dose (RP3D) High Dose Q2W

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled Phase IIb/III clinical trial aimed at evaluating the efficacy, safety, pharmacokinetics (PK), and immunogenicity profile of Efsubaglutide Alfa injection in overweight and obese subjects. The primary endpoint of the Phase IIb is the percentage change in body weight from baseline after 18 weeks of treatment. The primary endpoint of the Phase III is the percentage change in body weight from baseline after 30 weeks of treatment, the secondary endpoint is the percentage change in body weight from baseline after a cumulative 48 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the clinical study; fully understand and be informed about the study, and sign the informed consent form (ICF); willing to follow and capable of completing all study procedures.
2. Age ≥ 18 years (including the cutoff value, based on the time of signing the ICF), regardless of gender.
3. History of poor weight control through diet and exercise [defined as weight control failure if the subject has attempted at least 3 months of diet and exercise alone prior to screening without achieving a weight loss of ≥ 5.0% (based on subject self-report)].
4. Willing to follow the recommendations of the investigator regarding medication, diet, and exercise.
5. Stable weight within 3 months prior to screening (defined as a weight change < 5%, based on subject self-report).
6. Obesity: Body Mass Index (BMI) ≥ 28 kg/m² (including the cutoff value) with or without comorbidities; or overweight: BMI ≥ 24 and < 28 kg/m² with at least one weight-related comorbidity, including but not limited to prediabetes (impaired fasting glucose [FPG] and/or abnormal glucose tolerance), hypertension, dyslipidemia, non-alcoholic fatty liver disease, or obstructive sleep apnea syndrome.
7. Women of childbearing potential must have a negative blood pregnancy test during the screening period. Women of childbearing potential or male subjects and their partners must agree not to plan for pregnancy from the time of signing the ICF until 3 months after the last dose of the investigational drug, and voluntarily agree to use effective contraception, with no plans for sperm or egg donation.

Exclusion Criteria:

1. Allergic constitution or allergic to any component of the investigational drug.
2. Previously treated with Efsubaglutide Alfa injection.
3. Received glucagon-like peptide-1 (GLP-1) receptor agonists, dipeptidyl peptidase-4 (DPP-4) inhibitors, sodium-glucose co-transporter-2 (SGLT-2) inhibitors, insulin, metformin, insulin secretagogues, or thiazolidinediones (TZD) or any other weight-affecting anti-diabetic medication within the past 3 months before screening.
4. HbA1c ≥ 6.5% at screening, or previously diagnosed with Type 1 or Type 2 diabetes (based on the World Health Organization [WHO] 2020 diabetes diagnosis and classification standards).
5. History of severe hypoglycemia or recurrent symptomatic hypoglycemia (≥ 2 times in the past 6 months).
6. Known single-gene mutations, other diseases, or drug-induced obesity, including but not limited to hypothalamic obesity, pituitary obesity, hypothyroid obesity, Cushing's syndrome, insulinoma, growth hormone deficiency, acromegaly, pseudohypoparathyroidism, gonadal dysfunction, etc.
7. Clinically significant gastric emptying abnormalities (e.g., gastric outlet obstruction), severe chronic gastrointestinal diseases (e.g., active ulcers in the past 6 months), long-term use of drugs directly affecting gastrointestinal motility (including but not limited to mosapride, cisapride, etc.), or having undergone gastrointestinal surgery within the past 6 months and deemed unsuitable for participation by the investigator.
8. Use of weight-affecting medications within 3 months prior to screening, including tricyclic antidepressants, psychiatric medications, or sedative drugs (such as imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, sulpiride, clozapine, olanzapine, valproic acid, valproic acid derivatives, lithium salts, etc.). Note: Excluded if cumulative or continuous systemic steroid use is less than 14 days.
9. Use of non-prescription weight loss medications or appetite suppressants (including traditional Chinese medicine weight loss drugs) within 1 month prior to screening, or use of prescription weight loss medications (e.g., phentermine, sibutramine, orlistat) or lipid-dissolving injectables (e.g., lipolytic injections) within 3 months prior to screening.
10. Previously underwent weight-loss surgery (excluding acupuncture, liposuction, and abdominal fat removal within 1 year before screening), or plans to undergo surgery for obesity during the study period, such as gastric bypass surgery or gastric band surgery.
11. Currently on a weight loss plan and not in the maintenance phase.
12. History of hyperthyroidism or hypothyroidism, or thyroid-stimulating hormone (TSH) < 1×LLN (lower limit of normal) or TSH > 1.5×ULN (upper limit of normal).
13. Screening serum calcitonin ≥ 50 ng/L (or ≥ 50 pg/mL), or history of medullary thyroid cancer, multiple endocrine neoplasia (MEN) syndrome type 2A or 2B, or related family history (family history defined as a first-degree relative with the disease).
14. History of acute or chronic pancreatitis, cholecystectomy, or symptomatic gallbladder disease (patients with post-surgery resolved gallstones or cholecystectomy without sequelae can be enrolled), or known history of pancreatic injury or high-risk factors for pancreatitis, or screening with serum amylase or lipase > 2×ULN.
15. Any disease that could affect HbA1c measurement, such as hemolytic anemia, sickle cell disease, etc.
16. Currently receiving or have received chronic (> 14 days) systemic corticosteroid treatment in the past 3 months (excluding local, intraocular, intranasal, intra-articular, or inhaled formulations), or have evidence of severe, active autoimmune disorders (e.g., lupus or rheumatoid arthritis), and, in the opinion of the investigator, require or may require systemic corticosteroid treatment within the next 12 months.
17. History of malignancy within 5 years prior to screening, excluding clinically cured cervical carcinoma in situ, squamous cell carcinoma of the skin, or basal cell carcinoma within the past 5 years.
18. History of major surgery (e.g., thoracic, intracranial, or abdominal surgery) within 6 months prior to screening, or plans to undergo surgery that may affect study completion or adherence.
19. Meets any of the following cardiac function criteria: clinically significant arrhythmias or conduction abnormalities requiring clinical intervention; hereditary long QT syndrome or QTcF > 450 msec or currently taking medications that may prolong the QT interval or cause torsades de pointes; clinically significant cardiovascular diseases, including acute myocardial infarction, unstable angina, coronary artery bypass graft surgery, New York Heart Association (NYHA) class III or higher congestive heart failure, left ventricular ejection fraction (LVEF) < 50%, or uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg); other clinically significant cardiac abnormalities judged by the investigator.
20. History of hemorrhagic or ischemic stroke or transient ischemic attack within 6 months prior to screening.
21. Known infectious diseases: hepatitis B surface antigen (HBsAg) positive; hepatitis C virus (HCV) antibody positive and HCV RNA above the detection limit; human immunodeficiency virus (HIV) antibody positive; Treponema pallidum antibody positive.
22. Laboratory findings meeting any of the following: alanine aminotransferase (ALT) ≥ 3.0×ULN (subjects diagnosed with non-alcoholic fatty liver disease during screening and within the past 6 months with ALT ≤ 5.0×ULN may be enrolled); aspartate aminotransferase (AST) ≥ 3.0×ULN; total bilirubin (TBIL) ≥ 2.0×ULN; estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m² (CKD-EPI formula); fasting triglycerides (TG) > 5.65 mmol/L.
23. Known or suspected alcohol abuse within 1 year prior to screening (defined as male subjects consuming > 24 g alcohol per day, female subjects consuming > 12 g alcohol per day; 12 g alcohol is approximately equivalent to 300 mL beer, 100 mL wine, or 25 mL spirits).
24. Known or suspected drug abuse at screening.
25. Pregnant or breastfeeding women.
26. History of moderate to severe depression, anxiety, or serious mental disorders, such as schizophrenia, bipolar disorder, etc., or screening PHQ-9 score ≥ 15.
27. History of suicidal tendencies or suicide attempts.
28. Participation in a clinical trial involving vaccines, medical devices, or other drugs within 3 months prior to screening (except for observational studies).
29. The investigator or treating physician considers that the subject has any factors that may affect the evaluation of the efficacy or safety of the study, and is deemed unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1003 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight from baseline | Phase IIb (18 weeks) , Phase III (30 weeks)
Proportion of subjects with ≥5% reduction in body weight from baseline | Phase III (30 weeks)

SECONDARY OUTCOMES:
Proportion of subjects with ≥5% reduction in body weight from baseline | Phase IIb (18 weeks) , Phase III (48 weeks)
Proportion of subjects with ≥10%, and ≥15% reduction in body weight from baseline | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Percentage change in body weight from baseline | Phase III (48 weeks)
Change in body weight from baseline | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in BMI from baseline | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in waist circumference from baseline | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in hip circumference from baseline | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in blood pressure (diastolic and systolic) from baseline | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in lipid levels (triglycerides, total cholesterol, low-density lipoprotein cholesterol) from baseline, percentage change from baseline, and ratio to baseline. | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in blood glucose levels (FPG) from baseline | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in blood glucose levels (HbA1c) from baseline | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in blood glucose levels (fasting insulin) from baseline | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in blood glucose levels (insulin resistance index [HOMA-IR]) from baseline | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in blood uric acid levels from baseline | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in IWQOL-lite-CT (Impact of Weight on Quality of Life-Lite-Clinical Trial Version) Questionnaire Score from Baseline | Phase III (30 weeks and 48 weeks)

OTHER OUTCOMES:
Change in Total Body Fat Mass from Baseline Measured by Dual-Energy X-ray Absorptiometry | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in Liver Fat Content (LFC) from Baseline Measured by MRI-PDFF | Phase IIb (18 weeks) , Phase III (30 weeks and 48 weeks)
Change in Fibrosis-4 (FIB-4) Score from Baseline | Phase III (30 weeks and 48 weeks)
Change in Nonalcoholic Fatty Liver Disease Fibrosis Score (NFS) from Baseline | Phase III (30 weeks and 48 weeks)
Change in eGFR from Baseline | Phase III (30 weeks and 48 weeks)
Change in Urinary Albumin-to-Creatinine Ratio (ACR) from Baseline | Phase III (30 weeks and 48 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, M.D,Ph. D, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (41):
- China (41):
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Changzhou First People's Hospital, Changzhou
  - Sichuan Academy of Medical Sciences &Sichuan Provincial People's Hospital, Chengdu
  - Nanfang Hospital Southern Medical University, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliateo Hospital of Jinan University, Guangzhou
  - Zhujiang Hospital of Southern Medical University, Guangzhusi
  - The First People'S Hospital of Zunyi, Guizhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Henan University of Science and Technology, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Henan
  - Pingxiang People's Hospital, Jiangxi
  - Jincheng General Hospital, Jincheng
  - The Third Affiliated Hospital, Jinzhou
  - The First People's Hospital of Yunnan Province, Kunming
  - Luan City People's Hospital, Lu'an
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjing
  - Nan Jing First Hospital, Nanjing
  - The Second Hospital of Nanjing Medical University, Nanjing
  - The Affiliated Qingyuan Hospital ,Guangzhou Medical University（Qingyuan People's Hospital）, Qingyuan
  - The First Hospital of Qinhuangdao, Qinhuangdao
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Shandong
  - Shanghai Sixth People's Hospital Affiliated to Shanghai JiaoTong University, Shanghai
  - Shanghai General Hospital, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - The First Hospital Of China Medical University, Shenyang
  - Shenzhen Second People's Hospital, Shenzhen
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Suzhou Municipal Hospital, Suzhou
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - General Hospital of Tianjin Medical University, Tianjin
  - Tianjin Medical University Chu Hsien-I Memorial Hospital, Tianjin
  - Tenth People's Hospital Of Tongji University, Wuhan
  - Wuhan Third Hospital Tongren Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xianian
  - Yueyang Central Hospital, Yueyang

IPD SHARING:
Plan to Share IPD: No